CLINICAL TRIAL: NCT02251067
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel Group, Phase 2, Two-Part Adaptive Study to Evaluate the Safety and Efficacy of VPI-2690B Injection in Patients With Nephropathy Due to Diabetes
Brief Title: Phase 2 Study to Evaluate Safety & Efficacy of VPI-2690B in Diabetic Nephropathy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vascular Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VPI-CLIN-201-AD
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- VPI-2690B low dose (Active Comparator): 6 mg, VPI-2690B Injection, administered subcutaneously every 2 weeks for 48 weeks
  Interventions: Drug: VPI-2690B low dose
- VPI-2690B medium dose (Active Comparator): 18 mg, VPI-2690B Injection, administered subcutaneously every 2 weeks for 48 weeks
  Interventions: Drug: VPI-2690B medium dose
- Placebo (Placebo Comparator): 6 or 18 mg Placebo, administered subcutaneously every 2 weeks for 48 weeks
  Interventions: Drug: Placebo to match VPI-2690B
- VPI-2690B high dose (Active Comparator): 48 mg, VPI-2690B Injection, administered subcutaneously every 2 weeks for 48 weeks
  Interventions: Drug: VPI-2690B high dose

INTERVENTIONS:
Drug: VPI-2690B low dose — Comparison of different doses of study drug
  Arms: VPI-2690B low dose
Drug: VPI-2690B medium dose — Comparison of different doses of study drug
  Arms: VPI-2690B medium dose
Drug: Placebo to match VPI-2690B
  Arms: Placebo
Drug: VPI-2690B high dose — Comparison of different doses of study drug
  Arms: VPI-2690B high dose

SUMMARY:
The purpose of this study is to determine whether VPI-2690B Injection is effective in the treatment of diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* documented diabetic nephropathy in patients with either Type 1 or Type 2 diabetics
* HbA1c of 7.5-10.5%
* eGFR 30-110 mL/min/1.73m2
* stable ACEi/ARB dose regimen
* stable blood pressure
* BMI less than or equal to 45 kg/m2

Exclusion Criteria:

* non-diabetic renal disease
* history of solid organ or islet cell transplant
* history of malignancy within previous 5 years
* systemic immunosuppression therapy
* clinically significant liver disease, hepatitis B or C or HIV
* monoclonal antibody treatment within previous year
* recent acute renal injury or major surgery
* significant, recent body weight change
* biopsy proven glomerular disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in albuminuria | 50 weeks

SECONDARY OUTCOMES:
Change from baseline in eGFR | 50 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vascular Pharmaceuticals Inc Clinical Trial, Study Director — Vascular Pharmaceuticals, Inc.
Locations (34):
- United States (32):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - La Mesa, California
  - Riverside, California
  - Sacramento, California
  - Tustin, California
  - Cooper City, Florida
  - Coral Springs, Florida
  - Hialeah, Florida
  - Miami, Florida
  - St. Petersburg, Florida
  - Winter Park, Florida
  - Columbus, Georgia
  - Idaho Falls, Idaho
  - Mount Prospect, Illinois
  - Peoria, Illinois
  - Merrillville, Indiana
  - Boston, Massachusetts
  - Flint, Michigan
  - Kansas City, Missouri
  - Las Vegas, Nevada
  - Albany, New York
  - Asheville, North Carolina
  - Greenville, North Carolina
  - Morehead City, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Wooster, Ohio
  - Allentown, Pennsylvania
  - Nashville, Tennessee
  - El Paso, Texas
  - San Antonio, Texas
- Puerto Rico (2):
  - Ponce
  - San Juan